CLINICAL TRIAL: NCT01930500
Title: The Effectiveness of Neuropsychological Rehabilitation in Young Dyslexic Adults - a Single Blind, Randomized, Controlled Study
Brief Title: The Effectiveness of Neuropsychological Rehabilitation in Young Dyslexic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation Foundation, Finland (Other)
Collaborators: Helsinki University Central Hospital (Other); Social Insurance Institution, Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Luki-40211
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual neuropsychological rehabilitation (Experimental): 12 times 90 minutes, once per week or once per two weeks, during 5 months
  Interventions: Behavioral: Individual neuropsychological rehabilitation
- Group based neuropsychological rehabilitation (Experimental): 12 times 120 minutes + a brake, once per week or once per two weeks, during 5 months
  Interventions: Behavioral: Group based neuropsychological rehabilitation
- Control group (No Intervention): Control group does not receive neuropsychological rehabilitation or any other intervention during the first 5 months. After the control period they will be randomized to receive either individual or group based rehabilitation.

INTERVENTIONS:
Behavioral: Individual neuropsychological rehabilitation — Psychoeducation, teaching compensatory strategies and offering psychological support to better cope with dyslexia
  Arms: Individual neuropsychological rehabilitation
Behavioral: Group based neuropsychological rehabilitation — Psychoeducation, teaching compensatory strategies and offering psychological support and peer support to better cope with dyslexia
  Arms: Group based neuropsychological rehabilitation

SUMMARY:
The purpose of this study is to determine whether individual and/ group based neuropsychological rehabilitation focused on psychoeducation and teaching compensatory strategies has positive effects on the psychosocial wellbeing and perceived cognitive deficits in dyslexic young adults. The hypothesis is that both individual and group based neuropsychological rehabilitation show positive effects on the psychosocial wellbeing and perceived cognitive deficits. Another purpose of this study is to evaluate weather individual and group based neuropsychological rehabilitation have different kind of effects on the wellbeing of the participants and weather either one of the rehabilitation formats is more effective than the other.

DETAILED DESCRIPTION:
Background: Untreated dyslexia causes problems for individuals in studies, work and employment. High quality research on the best and most cost-effective rehabilitation methods is needed.

Objective: To study whether neuropsychological rehabilitation improves the psychosocial wellbeing and perceived cognitive deficits in dyslexic young adults and to evaluate potential differences between individual and group based neuropsychological rehabilitation.

Methods: Altogether 120 young adults diagnosed with dyslexia are randomized either to one of the intervention groups (individual neuropsychological rehabilitation / group neuropsychological rehabilitation) or to a control group which will receive either one of the interventions after a 5 month waiting period. All the study subjects are assessed with a short neuropsychological test battery as well as self-rating questionnaires evaluating mood, QoL, perceived cognitive deficits, and the impact of the learning disability at baseline, after five months (immediately after interventions or control period) and after 10 months. After 20 months a shorter follow-up using only self-ratings will be done via mail. Subjects in the intervention groups are offered neuropsychological rehabilitation in 12 sessions conducted once a week or once in two weeks during five months. Subjects in the control group do not receive any intervention for the first five months.

Results: The effects of interventions on psychosocial wellbeing and perceived cognitive deficits are evaluated using appropriate statistical procedures and comparing the differences between the interventions groups and the control group.

The present status: All the interventions are completed, follow-up data is still beeing collected

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of dyslexia
* age 18-35
* problems in studies, work or employment relating to dyslexia
* subjective and objective need for rehabilitation
* the native language is Finnish

Exclusion Criteria:

* other neurological condition than dyslexia
* other learning disabilities than dyslexia
* overall weak cognitive capacity
* psychiatric diagnosis
* severe depression
* alcohol or drug abuse
* neuropsychological rehabilitation received at the age of 16 or later

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Subjective cognitive performance | 5 months
  The effects of rehabilitation on subjective cognitive performance: Everyday Memory Questionnaire (EMQ)
Subjective reading related performance | 5 months
  Effects of rehabilitation on subjective reading related performance: Adult Reading History Questionnaire (ARHQ) modified

SECONDARY OUTCOMES:
Verbal fluency and executive control | 5 months
  These cognitive skills are measured using verbal fluency with category switching, Delis-Kaplan Executive Function System; D-KEFS. The score is the total number of correct words generated by the participant within the one-minute time-limit. The range for points is from 0 to as many words as can be generated by the rules within one minute. More points equals a better result.
Goal achievement | 5 months
  Goal achievement is measures using Goal Attainment Scaling (GAS). The attained goals set at the beginning of the intervention and measured on a scale from -2 to +2 at the end of the intervention. The score is based on a discussion with the therapist and the participant. A score below zero means that the set goal has not been reached. A score of 0 means that the goal has been reached and scores above 0 mean that the goal was reached over expectations.
Quality of life: QOLIBRI-OS | 5 months
  The effects of rehabilitation on quality of life are measured using the Quality of Life after Brain Injury Overall Scale (QOLIBRI-OS). The score ranges from 6-30. More points equals a better quality of life.
Mood | 5 months
  The effects of rehabilitation on mood are measured using Profile of Mood States (POMS). The Finnish version contains 38 questions and the total score ranges from 0 to 152. Less points means a better situation for mood.
Social and cognitive behavioral strategies | 5 months
  Strategy and Attribution Questionnaire (SAQ) bref consists of 20 questions using a 7-point-scale (from 1 = "strongly disagree" to 7 = "strongly agree") to assess social and cognitive behavioral strategies.
Processing speed and attention | 5 months
  These cognitive skills are measured using Symbol Digit Modalities test. The score ranges from 0 to 110. More points equals a better result.
Verbal learning | 5 months
  Verbal learning is measured using Word lists subtest (Wechsler Memory Test-III, WMS-III). The total score is between 0 - 48. More points equals a better result.
Reading comprehension | 5 months
  Reading comprehension is measured using V3, a part of a Finnish Ability Test Battery, "Kykytestistö AVO-9". The score ranges fron 0 to 20. More points equals a better result.
Visual fluency and executive control | 5 months
  These cognitive skills are measured using design fluency, Delis-Kaplan Executive Function System; D-KEFS. The score is the total number of correct drawings produced within a minute added togehter from three different one-minute long sessions with different rules. The range for points is from 0 to as many drawings as can be generated by the rules within the three one-minute sessions. More points equals a better result.
Working memory | 5 months
  Working memory is assesed using Digit span sequencing (Wechsler Adult Intelligence Scale - Fourth Edition, WAIS-IV). The total score is between 0 - 16. More points equals better result.

CONTACTS AND LOCATIONS:
Overall Officials: Erja Poutiainen, PhD, Study Director — Rehabilitation Foundation; Johanna Nukari, LicPsych, Principal Investigator — Rehabilitation Foundation
Locations (1):
- Rehabilitation Foundation, Helsinki, Malminkartano, Finland